CLINICAL TRIAL: NCT04320082
Title: Alteration of Blood-Brain-Barrier Permeability at Loss of Consciousness in Delirious Patients Recorded With Direct-Current Electroencephalography (ACDC)
Status: Terminated | Type: Observational
Why Stopped: The study staff has left the clinic.
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Ansthesiology and Operative Intensive Care Medicine, Charité - Universitätsmedizin Berlin, Charite University, Berlin, Germany
Other Study IDs: ACDC
Record Dates: First submitted 2020-03-23; First posted 2020-03-24 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elderly cohort: Patients >70 undergoing elective orthopaedic or trauma surgery under general anaesthesia.
- Young cohort: Patients between 18 and 30 undergoing elective orthopaedic or trauma surgery under general anaesthesia.

SUMMARY:
With this trial we aim to characterize the intraoperative signatures of the Direct-Current-Electroencephalogram (DC-EEG) of elderly patients developing a PostOperative Delirium (POD) compared to patients who do not develop a POD. We hereby intend to gain a better understanding of the electrical potential at the blood-brain-barrier (measured with DC-EEG) during general anaesthesia. Second, we want to study the effect of age on the DC-EEG by comparing a younger (18-30y) to an elderly cohort (>70). Third, we aim to couple the DC-EEG signatures to blood sample analysis in order to understand the relationship between metabolic, inflammatory and vascular reaction with the intraoperative DC-EEG.

DETAILED DESCRIPTION:
In order to study the intraoperative DC-EEG signatures of elderly patients coupled with lab data to evaluate the role of the age-dependent blood-brain barrier (BBB) dysfunction in general anesthesia and its meaning in POD pathophysiology following protocol will be followed:

1. On the day of the surgery the 21 DC-EEG sintered Ag/AgCl (silver chloride) electrodes will be placed before the start of anesthesia following the 10-20-system.
2. The first blood sample will be collected via the routinely placed intravenous catheter.
3. During the induction of anesthesia special care will be given to the exact time of loss of consciousness (LOC), defined with the suppression of the lid closure reflex.
4. Markers will be set at important time points of the anesthetic care (Baseline, start of analgesia/anesthesia, LOC, intubation, beginning of surgical procedure, end of anesthesia, regain of consciousness, extubation, admission recovery room).
5. Shortly after consciousness has vanished (5-10 minutes), a second blood sample will be drawn.
6. The DC-EEG recording will last until one hour after arrival at the recovery room, during which NuDesc score will be assessed every 15 minutes.
7. A third blood sample is to be collected in the recovery room. In the five days following surgery patients will be visited in the morning and in the evening to screen delirious symptoms with the help of standardized scores (NuDesc, DSM V, DDS). If patients are staying on the intensive care unit the CAM-ICU will be used.

Blood sample analysis will include blood cells count, electrolytes, inflammatory markers, cholesterols, proteins, structural BBB markers and markers of neuronal damage.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >70 years OR between 18 and 30
* Planned operation time >1 hour
* Expected hospital treatment period of 5 days,
* Anesthesia induction, anesthesia maintenance with either Propofol or an inhalative anesthetic agent as Sevoflurane or Desflurane,
* The ability to give informed consent

Exclusion Criteria:

* Age under 18 or between 31 and 69
* Patients with a history of neurological or psychiatric disorders
* Planned neurosurgery
* Current medication of tranquilizers / antidepressants
* Isolation of patients with multi-resistant Bacteria
* Inability of the patients to speak and/or read German
* Intraoperative use of ketamine, N²O, Etomidate or Dexmedetomidine
* Participation in a prospective interventional trial

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly Cohort: Patients >70 undergoing elective orthopaedic or trauma surgery under general anaesthesia.
  Young cohort: Patients between 18 and 30 undergoing elective orthopaedic or trauma surgery under general anaesthesia.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
1. DC-Shift (µV/sec) in the perioperative DC-EEG. | From the beginning of general anaesthesia to one hour after regain of consciousness
  Full-brain DC-EEG with 21 electrodes placed preoperatively following the 10/20-System and recording until one hour after regain of consciousness.

SECONDARY OUTCOMES:
Incidence of Postoperative Delirium | Patients will be follow until hospital discharge, or maximal until postoperative day 5
  Postoperative Delirium is defined according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V) and/or as ≥ 2 cumulative points in the nursing Delirium Screening Scale (Nu-DESC) and/or a positive Confusion Assessment Method (CAM) and/or Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) score and/or patient chart review that shows descriptions of Delirium.
Additional perioperative DC-EEG signatures: morphology, polarity (positive/negative), amplitude (µV) | From the beginning of general anaesthesia to one hour after regain of consciousness
  Full-brain DC-EEG with 21 electrodes placed preoperatively following the 10/20-System and recording until one hour after regain of Consciousness.
DC-EEG signatures in young (18-30) vs. elderly (>70) patients | From the beginning of general anaesthesia to one hour after regain of consciousness
  Full-brain DC-EEG with 21 electrodes placed preoperatively following the 10/20-System and recording until one hour after regain of consciousness
Analysis of pre-, intra- and postoperative blood parameters | : From shortly before the beginning of general anaesthesia to maximum one hour after arrival in the recovery room
  Blood samples will be drawn before the start of general anesthesia, shortly after loss of consciousness and in the recovery room.
Peri-operative, full-brain overall EEG band power | Up to the end of stay in the recovery room
  Full-brain EEG recording with surface Ag/AgCl electrodes Spectral analysis by Matlab Code/Lab Chart
Burst suppression duration | During anesthesia procedure
  Full-brain EEG recording with surface electrodes, raw EEG analysis
Duration of Delirium | Participants will be followed for the duration of hospital stay, or maximal until postoperative day 5
  Diagnostic and Statistical Manual of Mental Disorders (DSM-V); Nursing Delirium Screening Scale (Nu-DESC), Confusion Assessment Method for the Intensive Care Unit (CAM-ICU), Confusion Assessment Method (CAM), Chart Review
Intensive care unit length of stay | Participants will be followed for the duration of intensive care unit stay, an expected average of 5 days
  The stay is measured in days.
Hospital length of stay | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  The stay is measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany